CLINICAL TRIAL: NCT03517111
Title: Multi-level Effects of a Parenting Intervention for Enhancing Latino Youth Health Behaviors
Brief Title: The Impact of a Parenting Intervention on Latino Youth Health Behaviors
Acronym: FPNG+
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to interact with participants for intervention or data collection due to COVID-19 quarantine and social distancing restrictions.
Sponsor: Arizona State University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Sonia Vega-Lopez, Associate Professor, School of Nutrition and Health Promotion, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ASU6797; 2U54MD002316-11 (NIH)
Record Dates: First submitted 2018-03-22; First posted 2018-05-07 (Actual); Results first posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Diet Modification; Substance Use Disorders; Diabetes Mellitus Risk; Cardiovascular Risk Factor; Lifestyle Risk Reduction; Parenting
MeSH Terms: conditions — Substance-Related Disorders; Risk Reduction Behavior | interventions — Nutritional Status

STUDY DESIGN:
Intervention Model Description: Randomization to treatment conditions (FPNG+, FPNG, or comparison [RAD]) will occur at the school level. From the 18 participating schools, 6 each will be randomized into one of the three conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nutrition/substance use prevention (Experimental): Parenting and nutrition curriculum targeting substance use prevention and diet improvement.
  Interventions: Behavioral: Nutrition/substance use prevention
- Substance use prevention only (Active Comparator): Parenting curriculum targeting substance use prevention only.
  Interventions: Behavioral: Substance use prevention only
- Academic success program (Sham Comparator): Control program focused only on academic success.
  Interventions: Behavioral: Academic success program

INTERVENTIONS:
Behavioral: Nutrition/substance use prevention — Parenting program focusing on diet improvement and substance use prevention
  Other Names: FPNG+
  Arms: Nutrition/substance use prevention
Behavioral: Substance use prevention only — Parenting program focusing only on substance use prevention
  Other Names: FPNG
  Arms: Substance use prevention only
Behavioral: Academic success program — Program focusing on academic success and college acceptance
  Other Names: Realizing the American Dream (RAD)
  Arms: Academic success program

SUMMARY:
The purpose of this study is to test if a parenting program can be used to prevent substance use among Latino youth and at the same time promote healthy eating. Pairs of 7th grade students and one of their parents will be enrolled in the study and randomly assigned to three groups: an existing parenting intervention focusing on substance use prevention (FPNG), the enhanced parenting intervention that also has nutrition content (FPNG+), and a comparison program focused on academic success. Only parents will attend intervention sessions. Data will be collected from the parent and their 7th grade student to see how these programs impacted substance use, nutrition, and parenting. The investigators hypothesize that families receiving the FPNG+ will have improved nutrition habits than the other conditions. Students in both FPNG and FPNG+ will have lower substance use rates as compared to the academic success program. In addition, the effects of parenting strategies and sociocultural factors on the FPNG and FPNG+ results will be studied.

DETAILED DESCRIPTION:
Latino youth are a population at risk for chronic diseases because of their growing overweight and obesity rates, lack of adherence to nutrition and physical activity recommendations, and greater rates of tobacco, alcohol and other drugs use than youth of other ethnic groups. Parents are an important agent of change for youth due to their ability to create a home environment that promotes healthful behaviors (including substance use prevention and healthy nutrition), and parents' role as providers of resources to the family (including food). Parenting interventions are efficacious in preventing substance use among Latino youth, but few studies have used a family approach to promote healthy nutrition. Thus, the overall objective of the proposed project is to extend the scope of Families Preparing the New Generation (FPNG), an existing parenting program proven to help reduce substance use among Latino youth, to also promote healthy nutrition. The eco-developmental perspective will provide the theoretical foundation for the project for investigating risk and resiliency in Latino youth's drug use and nutrition behaviors. The main aims of the study are to (1) test the effects of a nutrition-enhanced parenting program (FPNG+) on substance use and nutrition among Latino youth, (2) explore how enhancing parenting skills impact the effects of the enhanced intervention, and (3) understand how social and cultural factors impact how the enhanced program works. The research team will first seek input from community members to create a nutrition-enhanced program that is acceptable to Latino parents of middle school students. The investigators will then collaborate with the American Dream Academy (ADA), an organization delivering an academic success program to families within middle schools throughout the Phoenix Area, to recruit 1,494 families who have a student in 7th grade to participate in the study. Parents from different schools will be offered one of three 10-week programs (assigned to each individual school): FPNG+ (substance use prevention and healthy nutrition), FPNG (substance use prevention only), and the ADA comparison program (focusing on academic success). Data will be collected from the 7th grade student and his/her participating parent before the start of the program, immediately after it ends, and 16 weeks later, to compare how the programs affect nutrition, substance use, and parenting. In a subgroup of 126 families (42 from each program), investigators will explore how the FPNG+ program affects diabetes and cardiovascular risk factors and whether the program induces changes in the types of foods available at participants' homes. For this, investigators will collect capillary blood samples from participants to measure glycosylated hemoglobin (a marker of diabetes risk) and cholesterol (a marker of cardiovascular risk), and blood pressure, as well as a list of foods that participants have at home. The long-term goal is to design and disseminate programs that contribute to helping parents assist their adolescent children develop and maintain long-lasting positive lifestyle behaviors in order to prevent substance use and chronic diseases.

ELIGIBILITY:
Inclusion criteria:

* Youth: ages 12-14
* Youth: Enrolled in 6th,7th, or 8th grade at the time of recruitment from the American Dream Academy (ADA) programs
* Adults: Age 18 or older
* Adults: Parent/caregiver/guardian of an eligible youth

Exclusion Criteria: None

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 844 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio F Marsiglia, PhD, Principal Investigator — Southwest Interdisciplinary Research Center, Arizona State University
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

REFERENCES:
- [Background] Vega-Lopez S, Marsiglia FF, Ayers S, Williams LR, Bruening M, Gonzalvez A, Vega-Luna B, Perilla A, Harthun M, Shaibi GQ, Delgado F, Rosario C, Hartmann L. Methods and rationale to assess the efficacy of a parenting intervention targeting diet improvement and substance use prevention among Latinx adolescents. Contemp Clin Trials. 2020 Feb;89:105914. doi: 10.1016/j.cct.2019.105914. Epub 2019 Dec 13. PMID 31843638
- [Background] Mercado M, Vega-Lopez S, Gonzalvez A, Vega-Luna B, Hoyt S, Martinez G, Ayers S, Marsiglia FF. Adaptation process of a culturally congruent parenting intervention for parents of Hispanic adolescents to an online synchronous format. Transl Behav Med. 2023 Apr 3;13(3):160-167. doi: 10.1093/tbm/ibac097. PMID 36617277
- [Result] Masek E, Gonzalvez A, Rankin L, Vega de Luna B, Valdez HJ, Hartmann L, Lorenzo E, Bruening M, Marsiglia FF, Harthun M, Vega-Lopez S. Qualitative Research on the Perceptions of Factors Influencing Diet and Eating Behaviors Among Primarily Latinx Seventh-Grade Students. J Acad Nutr Diet. 2023 Jul;123(7):1011-1021. doi: 10.1016/j.jand.2023.02.009. Epub 2023 Feb 14. PMID 36796757
- [Derived] Martinez GM, Vega-Lopez S, Ayers S, Gonzalvez A, Bruening M, Vega-Luna B, Marsiglia FF. Associations between parent-adolescent health-related conversations and mealtime media use among Hispanic families. Fam Syst Health. 2024 Jun;42(2):226-238. doi: 10.1037/fsh0000855. Epub 2023 Oct 23. PMID 37870808

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Goal was to enroll parent/6-8 grade age dyads;but some of the schools were grades K-8th grade.Per our community partner's terms, we opened up the study to all interested parents and did not turn anyone away.Parents whose child declined,or who had a child younger than the target age were still enrolled.These participants were not included in the final analyses,as they did not have a corresponding child.The numbers included in the participant flow are the total adults and children, not the dyads.
Units Other Than Participants: Schools
Period: Enrolled
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program
Started | 361; 6 Schools | 222; 5 Schools | 261; 5 Schools
Parents | 215; 6 Schools | 126; 5 Schools | 153; 5 Schools
Youth | 146; 6 Schools | 96; 5 Schools | 108; 5 Schools
Completed | 361; 6 Schools | 221; 5 Schools | 261; 5 Schools
Not Completed | 0; 0 Schools | 1; 0 Schools | 0; 0 Schools
Not completed — Withdrawal by Subject | 0 | 1 | 0
Period: T1 Survey (Week 0)
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program
Started | 361; 6 Schools | 221; 5 Schools | 261; 5 Schools
Parents | 132; 6 Schools | 125; 5 Schools | 153; 5 Schools
Youth | 101; 6 Schools | 96; 5 Schools | 108; 5 Schools
Completed | 361; 6 Schools | 221; 5 Schools | 261; 5 Schools
Not Completed | 0; 0 Schools | 0; 0 Schools | 0; 0 Schools
Period: T2 Survey (Week 10-12)
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program
Started | 361; 6 Schools | 221; 5 Schools | 261; 5 Schools
Parents | 132; 6 Schools | 71; 5 Schools | 98; 5 Schools
Youth | 101; 6 Schools | 57; 5 Schools | 76; 5 Schools
Completed | 233; 6 Schools | 128; 5 Schools | 174; 5 Schools
Not Completed | 128; 0 Schools | 93; 0 Schools | 87; 0 Schools
Not completed — Intervention workshops cancelled | 83 | 78 | 60
Not completed — Lost to Follow-up | 36 | 12 | 23
Not completed — Did not complete T2 survey, but continued with data collection | 9 | 3 | 4
Period: T3 Survey (Weeks 24-26)
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program
Started (Some participants skipped T2 survey, but completed T3) | 242; 6 Schools | 131; 5 Schools | 178; 5 Schools
Parents | 119; 6 Schools | 70; 5 Schools | 92; 5 Schools
Youth | 96; 6 Schools | 55; 5 Schools | 71; 5 Schools
Completed | 215; 6 Schools | 125; 5 Schools | 163; 5 Schools
Not Completed | 27; 0 Schools | 6; 0 Schools | 15; 0 Schools
Not completed — Lost to Follow-up | 27 | 6 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | Total
Number analyzed (Participants) | 361 | 221 | 261 | 843
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Parents and youth are entered and analyzed separately.
  years
    Parents: number analyzed (Participants) | 215 | 125 | 153 | 493
    Parents | 39.7 (6.913) | 40.48 (6.937) | 40.01 (6.894) | 39.99 (6.906)
    Youth: number analyzed (Participants) | 146 | 96 | 108 | 350
    Youth | 12.46 (.825) | 12.48 (1.02) | 12.35 (.9) | 12.44 (.903)
Sex: Female, Male [Count of Participants; unit: Participants]
  Parents: Female | 251 | 162 | 187 | 600
  Parents: Male | 110 | 59 | 74 | 243
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Parents and youth: Hispanic or Latino | 345 | 210 | 249 | 804
  Parents and youth: American Indian/Native American | 1 | 1 | 3 | 5
  Parents and youth: African American/Black | 1 | 1 | 0 | 2
  Parents and youth: Asian/Pacific Islander | 2 | 0 | 0 | 2
  Parents and youth: More than one category | 4 | 5 | 5 | 14
  Parents and youth: Unknown | 7 | 3 | 2 | 12
  Parents and youth: White or Anglo | 1 | 1 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 361 | 221 | 261 | 843
Adolescent Alcohol Use Frequency [Mean (Standard Deviation); unit: units on a scale] — Question: In the past 30 days, how many times have you...drunk more than a sip of beer, wine or liquor? Scale: 0 = 0; 1 = 1-2 times; 2 = 3-5 times; 3 = 6-9 times; 4 = 10-19 times; 5 = 20-39 times; 6 = 40 or more times Population: Analysis only conducted among adolescent participants.
  units on a scale
    number analyzed (Participants) | 143 | 95 | 107 | 345
    (all) | 0.05 (0.25) | 0.14 (0.66) | 0.10 (0.41) | 0.09 (0.445)
Adolescent Alcohol Use Amount (past 30 days) [Mean (Standard Deviation); unit: units on a scale] — Question: How many drinks of alcohol (more than a sip of beer, wine, or liquor) have you had in the past 30 days?
  Scale: 0=none; 1=one drink; 2=2-3 drinks; 3=4-7 drinks; 4=8-15 drinks; 5=16-30 drinks; 6=more than 30 drinks Population: Only adolescent participants were included in this analysis.
  units on a scale
    number analyzed (Participants) | 145 | 96 | 107 | 348
    (all) | 0.01 (0.08) | 0.11 (0.56) | 0.12 (0.54) | 0.07 (0.427)
Parent predicted intake of whole grains [Mean (Standard Deviation); unit: Ounce equivalents per day] — Primary dietary outcome - calculated from the Dietary Screener Questionnaire Population: Only parent participants were included in this analysis
  Ounce equivalents per day
    number analyzed (Participants) | 170 | 103 | 126 | 399
    (all) | 0.750 (0.335) | 0.694 (0.254) | 0.806 (0.618) | 0.753 (0.431)
Parent predicted intake of total added sugars [Mean (Standard Deviation); unit: Tsp equivalents per day] — Primary dietary outcome - calculated from the Dietary Screener Questionnaire Population: Only adult participants were included in this analysis.
  Tsp equivalents per day
    number analyzed (Participants) | 166 | 100 | 122 | 388
    (all) | 16.95 (6.90) | 16.14 (6.39) | 16.36 (6.26) | 16.56 (6.57)
Parent predicted intake of fruit and vegetables (including legumes) [Mean (Standard Deviation); unit: Cup equivalents per day] — Primary dietary outcome - calculated from the Dietary Screener Questionnaire Population: Only adult participants were included in this analysis
  Cup equivalents per day
    number analyzed (Participants) | 166 | 103 | 135 | 404
    (all) | 2.61 (0.80) | 2.50 (0.79) | 2.63 (0.74) | 2.59 (0.78)

OUTCOME MEASURES:

1. Primary Outcome: Adolescent Recent Alcohol Intake Frequency
Description: Question: In the past 30 days, how many times have you...drunk more than a sip of beer, wine or liquor? Scale: 0 = 0; 1 = 1-2 times; 2 = 3-5 times; 3 = 6-9 times; 4 = 10-19 times; 5 = 20-39 times; 6 = 40 or more times
Time Frame: (T1) Week 0, (T2) Week 10-12, (T3) Week 24-26
Population: Only adolescent participants were included in the analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program
Number analyzed (Participants) | 143 | 95 | 107
score on a scale
  T1 (Week 0) | 0.05 (0.25) | 0.14 (0.66) | 0.1 (0.41)
  T2 (Weeks 10-12): number analyzed (Participants) | 100 | 57 | 75
  T2 (Weeks 10-12) | 0.06 (0.28) | 0.18 (0.83) | 0.05 (0.23)
  T3 (Weeks 24-26): number analyzed (Participants) | 95 | 52 | 70
  T3 (Weeks 24-26) | 0.03 (0.18) | 0.12 (0.83) | 0.09 (0.41)

2. Primary Outcome: Adolescent Recent Alcohol Intake Amount
Description: Question: How many drinks of alcohol (more than a sip of beer, wine, or liquor) have you had in the past 30 days? Scale: 0 = None; 1 = One drink; 2 = 2-3 drinks; 3 = 4-7 drinks; 4=8-15 drinks; 5=16-30 drinks; 6= More than 30 drinks
Time Frame: (T1) Week 0, (T2) Week 10-12, (T3) Week 24-26
Population: Only adolescent participants were included in the analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program
Number analyzed (Participants) | 145 | 96 | 107
score on a scale
  T1 (Week 0) | 0.01 (0.08) | 0.11 (0.56) | 0.12 (0.54)
  T2 (Weeks 10-12): number analyzed (Participants) | 99 | 56 | 76
  T2 (Weeks 10-12) | 0.00 (0.00) | 0.14 (0.82) | 0.05 (0.23)
  T3 (Weeks 24-26): number analyzed (Participants) | 95 | 54 | 107
  T3 (Weeks 24-26) | 0.03 (0.18) | 0.11 (0.82) | 0.01 (0.12)

3. Primary Outcome: Drug Resistance Strategies
Description: Survey questions: Change in youths' responses to substance use offers in the past 30 days. Scale ranges from 0 (never responded in this way) to 5 (responded this way more than 10 times).
  Change in youths' intention to use substances measured as likely responses to hypothetical substance use offers. Scale ranges from 1 (Definitely no) to 4 (Definitely yes).
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Participants could skip questions; additionally, some participants didn't complete all three waves of data collection.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- All Conditions: All participants
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Conditions
Number analyzed (Participants) | 106 | 55 | 78 | 239
score on a scale
  Baseline (T1) drug resistance strategies: number analyzed (Participants) | 103 | 55 | 77 | 235
  Baseline (T1) drug resistance strategies | 1.1157 (1.43786) | 1.3364 (1.78485) | 1.2695 (1.5919) | 1.2177 (1.57104)
  T2 drug resistance strategies: number analyzed (Participants) | 98 | 55 | 76 | 229
  T2 drug resistance strategies | .7321 (1.11529) | .9273 (1.50745) | 1.1853 (1.79173) | .9294 (1.47036)
  T3 drug resistance strategies: number analyzed (Participants) | 91 | 51 | 69 | 211
  T3 drug resistance strategies | .7445 (1.34628) | .9314 (1.68751) | .7874 (1.49095) | .8037 (1.47654)
  Baseline (T1) intentions to use substances (higher score=higher intention): number analyzed (Participants) | 103 | 55 | 77 | 235
  Baseline (T1) intentions to use substances (higher score=higher intention) | 1.0947 (.25029) | 1.2045 (.44381) | 1.1526 (.96982) | 1.1394 (.34513)
  T2 intentions to use substances (higher score=higher intention): number analyzed (Participants) | 98 | 55 | 76 | 229
  T2 intentions to use substances (higher score=higher intention) | 1.1046 (.30865) | 1.1545 (.35516) | 1.1809 (.41553) | 1.1419 (.35825)
  T3 intentions to use substances (higher score=higher intention): number analyzed (Participants) | 93 | 53 | 69 | 215
  T3 intentions to use substances (higher score=higher intention) | 1.0914 (.25746) | 1.1179 (.30463) | 1.1739 (.50239) | 1.1244 (.36403)

4. Primary Outcome: Self-efficacy for Parenting Index
Description: A measure of parental beliefs that he/she is capable of performing parental roles/responsibilities
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: This outcome measure was removed from the survey, thus, there is no data to report.
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program
Number analyzed (Participants) | 0 | 0 | 0

5. Primary Outcome: Parents' Social Support
Description: Social Support Questionnaire score, scale from 1 to 7. Higher scores mean more social support.
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Participants could skip questions; additionally, some participants didn't complete all three waves of data collection.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- All Groups: Total for all three groups combined
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Groups
Number analyzed (Participants) | 106 | 55 | 78 | 239
score on a scale
  Baseline (T1) social support: number analyzed (Participants) | 105 | 55 | 78 | 238
  Baseline (T1) social support | 5.7689 (1.20103) | 5.4489 (1.51703) | 5.5684 (1.38217) | 5.6292 (1.33993)
  T2 social support: number analyzed (Participants) | 88 | 49 | 70 | 207
  T2 social support | 5.8381 (1.24913) | 5.6591 (1.38356) | 5.5846 (1.44316) | 5.71 (1.34744)
  T3 social support: number analyzed (Participants) | 85 | 51 | 66 | 202
  T3 social support | 5.7186 (1.1698) | 5.4725 (1.32787) | 5.5744 (1.28869) | 5.6094 (12.444)

6. Primary Outcome: Parent Self-agency
Description: Gauges the parent's sense of parenting competence and ability to positively influence the child's development. Scale from 1-5, with higher score=more agency.
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Participants could skip questions; additionally, not everyone completed all three waves of data collection.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Conditions
Number analyzed (Participants) | 106 | 55 | 78 | 239
score on a scale
  Baseline (T1) parental self agency | 4.221 (.51603) | 4.1176 (.55733) | 4.2744 (.51299) | 4.2146 (.52579)
  T2 parental self agency: number analyzed (Participants) | 87 | 49 | 70 | 206
  T2 parental self agency | 4.3879 (.51354) | 4.3868 (.46939) | 4.314 (.52859) | 4.3625 (.50744)
  T3 parental self agency: number analyzed (Participants) | 85 | 51 | 67 | 203
  T3 parental self agency | 4.3946 (.42518) | 4.4078 (.46167) | 4.3822 (.49498) | 4.3938 (.45615)

7. Primary Outcome: Overall Family Functioning- Parental Monitoring Subscale
Description: Survey questions (parents) measuring: Change in parental monitoring. Average of a 9-item scale, where each question is measured on a 5-point scale (1=Never, 5=Always).
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Participants could skip questions; additionally, not everyone completed all three waves of data collection.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Conditions
Number analyzed (Participants) | 106 | 55 | 78 | 239
score on a scale
  Baseline (T1) parental monitoring score (Week 0): number analyzed (Participants) | 79 | 32 | 35 | 146
  Baseline (T1) parental monitoring score (Week 0) | 4.288 (.48584) | 4.2471 (.47745) | 4.6252 (.41436) | 4.3599 (.48844)
  T2 parental monitoring score: number analyzed (Participants) | 88 | 49 | 69 | 206
  T2 parental monitoring score | 4.5216 (.47837) | 4.424 (.43793) | 4.5574 (.38802) | 4.5104 (.44107)
  T3 parental monitoring score: number analyzed (Participants) | 85 | 51 | 67 | 203
  T3 parental monitoring score | 4.5096 (.46168) | 4.4454 (.48924) | 4.5283 (.49091) | 4.4996 (.47716)

8. Primary Outcome: Overall Family Functioning- Parental Involvement
Description: From Gorman-Smith, Tolan, Zelli & Huesmann (1996) - These items measure the extent to which the parent is involved in the child's life. Respondents are asked to indicate how often they engage in certain interactions with their children (Q1-2) and how often the child is involved in family activities (Q3-10). For the first two questions, (when was the most recent time parent and youth talked about certain things), the scale goes from 1 (I don't know) to 5 (yesterday or today). For questions 3-10, activities include: how often the youth helps with family fun activities, how often parent and youth have a friendly talk, whether the youth helps with chores, or errands, etc. The scale goes from 1 (hardly ever) to 5 (often). Point values are summed (MIN=10, MAX=50), and then divided by the total number of items. Higher scores indicate greater levels of parental monitoring and involvement.
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Participants could skip questions; additionally, not everyone completed all three waves of data collection.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Conditions
Number analyzed (Participants) | 106 | 55 | 78 | 239
score on a scale
  Baseline (T1) parental involvement: number analyzed (Participants) | 106 | 54 | 78 | 238
  Baseline (T1) parental involvement | 4.178 (.54274) | 4.1796 (.56556) | 4.4319 (.49781) | 4.2616 (.54475)
  T2 parental involvement (Week 10-12): number analyzed (Participants) | 88 | 49 | 70 | 207
  T2 parental involvement (Week 10-12) | 4.437 (.4347) | 4.4277 (.36648) | 4.5902 (.40566) | 4.4866 (.41442)
  T3 parental involvement (Week 24-26): number analyzed (Participants) | 85 | 51 | 67 | 203
  T3 parental involvement (Week 24-26) | 4.2609 (.5196) | 4.3686 (.49051) | 4.4788 (.51803) | 4.3599 (.51801)

9. Primary Outcome: Overall Family Functioning- Family Support
Description: Survey questions (parents) measuring: Change in family support,
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Scale was removed from the final survey; there is no data to report.
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program
Number analyzed (Participants) | 0 | 0 | 0

10. Primary Outcome: Overall Family Functioning: Family Conflict
Description: Sub-scale measuring family conflict.
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Sub-scale was removed from survey. There is no data to report.
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program
Number analyzed (Participants) | 0 | 0 | 0

11. Primary Outcome: Overall Family Functioning- Familism
Description: Survey questions (parents) measuring familism subscale.
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Familism subscale was removed from final survey. There is no data to report.
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program
Number analyzed (Participants) | 0 | 0 | 0

12. Primary Outcome: Acculturation- Mexican Orientation Scale
Description: Acculturation Rating Scale for Mexican Americans-II (ARSMA-II) asks participants to indicate on a five point likert scale (Not at all (1) and Extremely often or almost always (5)) the extent to which they engage in certain cultural behaviors. The Mexican Orientation Subscale (MOS) consists of 17 Mexican oriented behaviors, which asks participants to indicate on the five point likert scale (Not at all (1) and Extremely often or almost always (5)) the extent to which they engage in Mexican-oriented behaviors. Means for each subscale are calculated, higher score indicates higher Mexican orientation.
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Parent results. Participants could skip questions. Additionally, some participants didn't complete all three waves of data collection.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Conditions
Number analyzed (Participants) | 106 | 55 | 78 | 239
score on a scale
  Baseline (T1) Mexican oriented scale (MOS)- Parents: number analyzed (Participants) | 105 | 55 | 77 | 237
  Baseline (T1) Mexican oriented scale (MOS)- Parents | 4.4314 (.57546) | 4.4418 (.55903) | 4.3171 (.78652) | 4.3967 (.64787)
  T2 Mexican oriented scale (MOS)- Parents: number analyzed (Participants) | 88 | 49 | 70 | 207
  T2 Mexican oriented scale (MOS)- Parents | 4.5019 (.50063) | 4.4905 (.55794) | 4.4905 (.68682) | 4.4953 (.58002)
  T3 Mexican oriented scale (MOS)- Parents: number analyzed (Participants) | 84 | 50 | 67 | 201
  T3 Mexican oriented scale (MOS)- Parents | 4.427 (.62828) | 4.5173 (.54901) | 4.502 (.703) | 4.4745 (.63436)

13. Primary Outcome: Acculturation- Anglo Orientation Subscale
Description: Acculturation Rating Scale for Mexican Americans-II (ARSMA-II) asks participants to indicate on a five point likert scale (Not at all (1) and Extremely often or almost always (5)) the extent to which they engage in certain cultural behaviors. The Anglo Orientation Subscale (AOS) consists of 13 items, which asks participants to indicate on the five point likert scale (Not at all (1) and Extremely often or almost always (5)) the extent to which they engage in Anglo oriented behaviors. Means for each subscale are calculated, higher score indicates higher Anglo orientation.
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Conditions
Number analyzed (Participants) | 106 | 55 | 78 | 239
score on a scale
  Baseline (T1) Anglo oriented scale (AOS)- Parents: number analyzed (Participants) | 102 | 51 | 77 | 230
  Baseline (T1) Anglo oriented scale (AOS)- Parents | 2.2827 (.85561) | 2.3876 (1.10831) | 2.3387 (1.05454) | 2.3247 (.98075)
  T2 Anglo oriented scale (AOS)- Parents: number analyzed (Participants) | 87 | 49 | 69 | 205
  T2 Anglo oriented scale (AOS)- Parents | 2.3149 (.86206) | 2.2714 (.96525) | 2.2906 (1.04594) | 2.2963 (.94736)
  T3 Anglo oriented scale (AOS)- Parents: number analyzed (Participants) | 84 | 51 | 63 | 198
  T3 Anglo oriented scale (AOS)- Parents | 2.3889 (.86462) | 2.3033 (.96986) | 2.4354 (1.10092) | 2.3816 (.96834)

14. Primary Outcome: Multidimensional Acculturative Stress Inventory
Description: Measures how often a person experienced certain acculturation situations and how stressful they were.
  Scale ranges from 0 (No, did not happen to me) to 5 (Extremely stressful). Mean score is created, where higher values indicate more acculturative stress.
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Parent results. Participants could skip questions; additionally, not all participants completed all data collection waves.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Conditions
Number analyzed (Participants) | 106 | 55 | 78 | 239
score on a scale
  Baseline (T1) acculturation stress | 1.783 (.7705) | 1.8831 (.81977) | 1.8571 (.78178) | 1.8302 (.78358)
  T2 acculturation stress: number analyzed (Participants) | 87 | 49 | 70 | 206
  T2 acculturation stress | 1.6521 (.67318) | 1.7172 (.70137) | 1.8738 (.88159) | 1.7429 (.75921)
  T3 acculturation stress: number analyzed (Participants) | 85 | 51 | 67 | 203
  T3 acculturation stress | 1.5235 (.62859) | 1.5014 (.63398) | 1.6951 (.85711) | 1.5746 (.71491)

15. Primary Outcome: Nutrition Outcomes- Fruit Intake
Description: NCI Dietary Screener: Change in intake of fruit- estimated cups per day
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Data was split up by parent and youth- they are reported separately.
Measure: Mean (Standard Deviation); unit: cups
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Conditions
Number analyzed (Participants) | 212 | 110 | 156 | 478
cups
  Baseline (T1) predicted intake of fruit per day (cup equivalents) - Parents: number analyzed (Participants) | 92 | 48 | 70 | 210
  Baseline (T1) predicted intake of fruit per day (cup equivalents) - Parents | 1.1578 (.64193) | 1.0087 (.34519) | 1.1194 (.55524) | 1.1109 (.55802)
  Baseline (T1) predicted intake of fruit per day (cup equivalents) - Youth: number analyzed (Participants) | 88 | 42 | 66 | 196
  Baseline (T1) predicted intake of fruit per day (cup equivalents) - Youth | .9929 (.55339) | 1.1968 (.77707) | 1.3499 (.94983) | 1.1568 (.76773)
  T2 predicted intake of fruit per day (cup equivalents) - Parents: number analyzed (Participants) | 74 | 41 | 62 | 177
  T2 predicted intake of fruit per day (cup equivalents) - Parents | 1.1115 (.52472) | .9861 (.42231) | 1.0496 (.64964) | 1.0608 (.55084)
  T2 predicted intake of fruit per day (cup equivalents) - Youth: number analyzed (Participants) | 75 | 41 | 57 | 173
  T2 predicted intake of fruit per day (cup equivalents) - Youth | 1.0778 (1.06928) | .9379 (.68743) | 1.0637 (.67436) | 1.04 (.86785)
  T3 predicted intake of fruit per day (cup equivalents) - Parents: number analyzed (Participants) | 81 | 50 | 65 | 196
  T3 predicted intake of fruit per day (cup equivalents) - Parents | .9626 (.41106) | .8214 (.23419) | .9511 (.37812) | .9227 (.3655)
  T3 predicted intake of fruit per day (cup equivalents) - Youth: number analyzed (Participants) | 89 | 51 | 64 | 204
  T3 predicted intake of fruit per day (cup equivalents) - Youth | .9062 (.52541) | .8979 (.46743) | .8071 (.37732) | .873 (.4687)

16. Primary Outcome: Nutrition Outcomes-vegetables
Description: NCI Dietary Screener: Change in intake of vegetables- estimated cups per day
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Data was split up by parent and youth- they are reported separately.
Measure: Mean (Standard Deviation); unit: cups
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Conditions
Number analyzed (Participants) | 212 | 110 | 156 | 478
cups
  Baseline (T1) predicted intake of vegetables per day (cup equivalents) - Parents: number analyzed (Participants) | 86 | 46 | 69 | 201
  Baseline (T1) predicted intake of vegetables per day (cup equivalents) - Parents | 1.5737 (.44437) | 1.5656 (.43126) | 1.6431 (.54488) | 1.5957 (.47739)
  Baseline (T1) predicted intake of vegetables per day (cup equivalents) - Youth: number analyzed (Participants) | 75 | 38 | 56 | 169
  Baseline (T1) predicted intake of vegetables per day (cup equivalents) - Youth | 1.1755 (.92976) | 1.0472 (.58324) | 1.105 (.67146) | 1.1233 (.77842)
  T2 predicted intake of vegetables per day (cup equivalents) - Parents: number analyzed (Participants) | 64 | 36 | 55 | 155
  T2 predicted intake of vegetables per day (cup equivalents) - Parents | 1.7107 (.56475) | 1.4978 (.38068) | 1.5468 (.34581) | 1.6031 (.46247)
  T2 predicted intake of vegetables per day (cup equivalents) - Youth: number analyzed (Participants) | 67 | 31 | 46 | 144
  T2 predicted intake of vegetables per day (cup equivalents) - Youth | 1.0538 (.6498) | .9821 (.27975) | .9756 (.39423) | 1.0134 (.51151)
  T3 predicted intake of vegetables per day (cup equivalents) - Parents: number analyzed (Participants) | 80 | 49 | 62 | 191
  T3 predicted intake of vegetables per day (cup equivalents) - Parents | 1.6077 (.43995) | 1.5163 (.39161) | 1.4687 (.3251) | 1.5391 (.3961)
  T3 predicted intake of vegetables per day (cup equivalents) - Youth: number analyzed (Participants) | 86 | 50 | 65 | 201
  T3 predicted intake of vegetables per day (cup equivalents) - Youth | 1.0941 (.47764) | .9209 (.32772) | .9903 (.35313) | 1.0175 (.41021)

17. Primary Outcome: Nutrition Outcomes-sugar-laden Foods
Description: NCI Dietary Screener: Change in intake of added sugars- estimated teaspoons per day
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Data was split up by parent and youth- they are reported separately.
Measure: Mean (Standard Deviation); unit: teaspooons
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Conditions
Number analyzed (Participants) | 212 | 110 | 156 | 478
teaspooons
  Baseline (T1) predicted intake of added sugars per day (tsp equivalents) - Parents: number analyzed (Participants) | 80 | 37 | 58 | 175
  Baseline (T1) predicted intake of added sugars per day (tsp equivalents) - Parents | 17.6583 (7.3443) | 15.9911 (5.10751) | 16.3719 (6.46963) | 16.8794 (6.6431)
  Baseline (T1) predicted intake of added sugars per day (tsp equivalents) - Youth: number analyzed (Participants) | 77 | 35 | 48 | 160
  Baseline (T1) predicted intake of added sugars per day (tsp equivalents) - Youth | 17.6124 (6.21487) | 18.4285 (5.61468) | 18.4825 (6.48959) | 18.052 (6.15085)
  T2 predicted intake of added sugars per day (tsp equivalents) - Parents: number analyzed (Participants) | 58 | 33 | 50 | 141
  T2 predicted intake of added sugars per day (tsp equivalents) - Parents | 14.5004 (4.14736) | 13.9483 (2.7104) | 16.2402 (6.42155) | 14.9881 (4.90186)
  T2 predicted intake of added sugars per day (tsp equivalents) - Youth: number analyzed (Participants) | 77 | 32 | 47 | 156
  T2 predicted intake of added sugars per day (tsp equivalents) - Youth | 17.702 (5.9984) | 16.5829 (3.42218) | 17.8928 (7.67179) | 17.5299 (6.13922)
  T3 predicted intake of added sugars per day (tsp equivalents) - Parents: number analyzed (Participants) | 80 | 51 | 61 | 192
  T3 predicted intake of added sugars per day (tsp equivalents) - Parents | 15.3366 (5.70302) | 14.3803 (4.26402) | 14.6353 (4.68844) | 14.8598 (5.02892)
  T3 predicted intake of added sugars per day (tsp equivalents) - Youth: number analyzed (Participants) | 91 | 50 | 67 | 208
  T3 predicted intake of added sugars per day (tsp equivalents) - Youth | 17.8769 (5.85852) | 16.4674 (4.52392) | 16.4405 (4.67735) | 17.0754 (5.21967)

18. Primary Outcome: Child Feeding Questionnaire- Weight-related Outcomes
Description: 3 item subscale measuring how often parents discussed certain weight-related topics with their adolescent (1=Never or rarely; 5=Almost every day).
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Participants could skip questions; additionally, not everyone completed all three waves of data collection.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Conditions
Number analyzed (Participants) | 106 | 55 | 78 | 239
score on a scale
  Baseline (T1) frequency of weight related topics | 2.6824 (1.28761) | 2.5879 (1.18411) | 2.4637 (1.26635) | 2.5893 (1.25596)
  T2 frequency of weight related topics: number analyzed (Participants) | 88 | 49 | 70 | 207
  T2 frequency of weight related topics | 2.8144 (1.34559) | 2.7619 (1.38109) | 2.6190 (1.33005) | 2.7359 (1.34503)
  T3 frequency of weight related topics: number analyzed (Participants) | 85 | 51 | 65 | 201
  T3 frequency of weight related topics | 2.6078 (1.32355) | 2.5294 (1.28958) | 2.5051 (1.28492) | 2.5547 (1.29692)

19. Primary Outcome: Child Feeding Questionnaire- Health-related Outcomes
Description: 3 item subscale measuring how often parents discussed certain health-related topics with their adolescent (1=Never or rarely; 5=Almost every day).
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Participants could skip questions; additionally, not everyone completed all three waves of data collection.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Conditions
Number analyzed (Participants) | 106 | 55 | 78 | 239
score on a scale
  Baseline (T1) frequency of health related topics: number analyzed (Participants) | 106 | 55 | 77 | 238
  Baseline (T1) frequency of health related topics | 3.9497 (.90477) | 4.0242 (.80086) | 4.1948 (.84872) | 4.0462 (.86675)
  T2 frequency of health related topics: number analyzed (Participants) | 88 | 49 | 70 | 207
  T2 frequency of health related topics | 4.2083 (.66343) | 4.2381 (.76980) | 4.2857 (.75349) | 4.2415 (.71782)
  T3 frequency of health related topics: number analyzed (Participants) | 85 | 51 | 67 | 203
  T3 frequency of health related topics | 4.0196 (.79074) | 4.0654 (.81927) | 4.1567 (.72873) | 4.0764 (.77665)

20. Primary Outcome: Food Insecurity
Description: This five-item scale is based on an 18-item validated food insecurity scale (Blumberg et al., 1999), for use when resources do not allow the use of the full scale. It assesses financially-based food insecurity and hunger in households with and without children. Questions 1 and 2 assess if food bought didn't last, and if they couldn't afford balanced meals; scale from 1=often true to 3=never true. The rest of the questions ask about actions the parent had to take due to lack of food; it's measured on a three-point scale where 1=No, 2=Yes, and 3=I don't know.
  The total number of affirmative responses is tallied: Questions 1 & 2, "Often" and "Sometimes" are considered affirmative responses; Question 3, "Yes, some months but not every month" and "Yes, almost every month" are considered affirmative responses; Questions 4 and 5, "Yes" is considered affirmative response. Minimum value is 0, maximum value is five. A greater score indicates higher level of food insecurity.
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Participants could skip questions; additionally, some participants didn't complete all three waves of data collection.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Conditions
Number analyzed (Participants) | 106 | 55 | 78 | 239
score on a scale
  Baseline (T1) food insecurity: number analyzed (Participants) | 104 | 54 | 77 | 235
  Baseline (T1) food insecurity | .6538 (1.13008) | .8704 (1.04694) | 1.1818 (1.44848) | .8766 (1.24279)
  T2 food insecurity: number analyzed (Participants) | 86 | 47 | 69 | 202
  T2 food insecurity | .6163 (1.1598) | .7872 (1.28429) | .9275 (1.45843) | .7634 (1.2979)
  T3 food insecurity: number analyzed (Participants) | 84 | 51 | 66 | 201
  T3 food insecurity | .7143 (1.14672) | .6078 (1.04074) | .9394 (1.41289) | .7612 (1.21766)

21. Secondary Outcome: Body Weight (kg)
Description: Measured body weight in kilograms (kg) for parents and youth. Calculated by taking the average of 3 consecutive weight readings.
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Only a subset of participants was selected for these additional home-based data collection measures. In-person data collection was halted due to the onset of the COVID-19 pandemic, hence sample sizes for T2 and T3 are small.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Conditions
Number analyzed (Participants) | 106 | 55 | 78 | 239
kg
  Baseline (T1) weight- Parents: number analyzed (Participants) | 26 | 17 | 29 | 72
  Baseline (T1) weight- Parents | 81.823 (19.075) | 83.292 (25.989) | 82.587 (18.0516) | 82.478 (20.2276)
  Baseline (T1) weight- Youth: number analyzed (Participants) | 25 | 17 | 29 | 71
  Baseline (T1) weight- Youth | 57.108 (13.7608) | 71.3135 (15.8803) | 58.6322 (14.26533) | 61.1343 (15.41305)
  T2 weight- Parents: number analyzed (Participants) | 20 | 16 | 27 | 63
  T2 weight- Parents | 80.9917 (15.62227) | 78.8146 (17.13268) | 80.3383 (14.52931) | 80.1587 (15.33090)
  T2 weight- Youth: number analyzed (Participants) | 20 | 16 | 26 | 62
  T2 weight- Youth | 58.9483 (14.02246) | 71.3521 (16.8629) | 59.9987 (14.81378) | 62.5898 (15.76246)
  T3 weight- Parents: number analyzed (Participants) | 15 | 13 | 23 | 51
  T3 weight- Parents | 82.7422 (17.53879) | 80.6408 (16.41642) | 81.1275 (14.31813) | 81.4784 (15.54774)
  T3 weight- Youth: number analyzed (Participants) | 14 | 12 | 22 | 48
  T3 weight- Youth | 56.3952 (12.9495) | 75.8417 (14.3459) | 61.1818 (15.6966) | 63.4507 (16.15782)

22. Secondary Outcome: Height
Description: Measured height for parents and youth in centimeters. Calculated by taking the average of three consecutive readings.
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Only a subset of participants was selected for this additional home-based data collection measure. In-person data collection was halted due to the onset of the COVID-19 pandemic, hence sample sizes for T2 and T3 are small.
Measure: Mean (Standard Deviation); unit: centimeters (cm.)
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Conditions
Number analyzed (Participants) | 106 | 55 | 78 | 239
centimeters (cm.)
  Baseline (T1) height- Parents: number analyzed (Participants) | 26 | 17 | 29 | 72
  Baseline (T1) height- Parents | 159.1526 (6.883) | 157.2784 (8.67363) | 158.7782 (7.64709) | 158.5593 (7.5656)
  Baseline (T1) height- Youth: number analyzed (Participants) | 25 | 17 | 29 | 71
  Baseline (T1) height- Youth | 156.3627 (7.80219) | 157.8647 (6.98786) | 157.9218 (7.1736) | 157.3592 (7.2914)
  T2 height- Parents: number analyzed (Participants) | 20 | 16 | 27 | 63
  T2 height- Parents | 159.435 (5.74194) | 156.8854 (8.85073) | 158.6642 (7.29788) | 158.4571 (7.2356)
  T2 height- Youth: number analyzed (Participants) | 20 | 16 | 26 | 62
  T2 height- Youth | 158.26 (8.34932) | 159.7792 (7.07612) | 159.6308 (7.3811) | 158.9688 (7.5309)
  T3 height- Parents: number analyzed (Participants) | 15 | 13 | 23 | 51
  T3 height- Parents | 158.4933 (6.4590) | 158.2562 (9.3633) | 157.9478 (7.23469) | 158.1869 (7.4705)
  T3 height- Youth: number analyzed (Participants) | 14 | 12 | 22 | 48
  T3 height- Youth | 158.931 (8.31398) | 158.7942 (7.17494) | 160.485 (8.22258) | 159.609 (7.8766)

23. Secondary Outcome: Body Mass Index for Parents
Description: Calculated BMI (body max index) for parents estimated by dividing weight (in kg) by height (in m) squared, with the unit of measure being kg/m^2. Typically, 18.5-24.9 is considered healthy weight; 25.0-29.9 is overweight; and equal or greater than 30.0 indicates obesity.
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Only a small subset of participants were selected for these biometric data collection procedures. In-person data collection was halted due to the onset of the COVID-19 pandemic, hence sample sizes for T2 and T3 are small.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Groups
Number analyzed (Participants) | 212 | 110 | 156 | 478
kg/m^2
  Baseline (T1) BMI- Parents: number analyzed (Participants) | 26 | 17 | 29 | 72
  Baseline (T1) BMI- Parents | 32.1158 (6.2109) | 33.5704 (9.6650) | 32.7239 (6.3371) | 32.7042 (7.12274)
  T2 BMI- Parents: number analyzed (Participants) | 20 | 16 | 27 | 63
  T2 BMI- Parents | 31.8463 (5.8633) | 32.1539 (7.8066) | 31.997 (5.8658) | 31.9889 (6.3025)
  T3 BMI- Parents: number analyzed (Participants) | 15 | 13 | 23 | 51
  T3 BMI- Parents | 32.8285 (6.12625) | 32.507 (8.3170) | 32.5999 (5.82704) | 32.6435 (6.4854)

24. Secondary Outcome: Systolic Blood Pressure
Description: Measured systolic blood pressure using an automated blood pressure monitor. Calculated by taking the average of three consecutive measures. Normal range is less than 120mm Hg (units of millimeters of mercury).
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Only a small subsample was selected to receive these additional data collection measures.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Groups
Number analyzed (Participants) | 212 | 110 | 156 | 478
mm Hg
  Baseline (T1) average systolic blood pressure- Parents: number analyzed (Participants) | 26 | 17 | 29 | 72
  Baseline (T1) average systolic blood pressure- Parents | 114.705 (16.9114) | 117.0 (15.4083) | 120.8851 (20.9567) | 117.7361 (18.3016)
  Baseline (T1) average systolic blood pressure- Youth: number analyzed (Participants) | 25 | 17 | 29 | 71
  Baseline (T1) average systolic blood pressure- Youth | 103.627 (11.6965) | 107.9804 (13.7742) | 102.6667 (10.8189) | 104.227 (11.9016)
  T2 average systolic blood pressure- Parents: number analyzed (Participants) | 20 | 16 | 27 | 63
  T2 average systolic blood pressure- Parents | 109.333 (9.0036) | 108.75 (15.8022) | 114.9753 (19.8397) | 111.6032 (16.0945)
  T2 average systolic blood pressure- Youth: number analyzed (Participants) | 20 | 16 | 26 | 62
  T2 average systolic blood pressure- Youth | 106.35 (11.922) | 106.0625 (10.6153) | 103.0513 (8.7405) | 104.8925 (10.2855)
  T3 average systolic blood pressure- Parents: number analyzed (Participants) | 15 | 13 | 23 | 51
  T3 average systolic blood pressure- Parents | 113.5333 (10.7959) | 116.2051 (12.2039) | 121.6812 (20.8684) | 117.8889 (16.5239)
  T3 average systolic blood pressure- Youth: number analyzed (Participants) | 14 | 12 | 22 | 48
  T3 average systolic blood pressure- Youth | 101.7143 (9.12483) | 105.5553 (7.9194) | 104.3939 (9.2127) | 103.9027 (8.8242)

25. Secondary Outcome: Diastolic Blood Pressure
Description: Measured diastolic blood pressure using an automated blood pressure monitor. Calculated by taking the average of three consecutive measures. Normal range is less than 80 mmHg (units of millimeters of mercury).
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Only a small subsample was selected for these biometric data collection.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Groups
Number analyzed (Participants) | 212 | 110 | 156 | 478
mm Hg
  Baseline (T1) average diastolic blood pressure - Parents: number analyzed (Participants) | 26 | 17 | 29 | 72
  Baseline (T1) average diastolic blood pressure - Parents | 71.667 (11.549) | 71.588 (10.725) | 75.7471 (11.539) | 73.2917 (11.3804)
  Baseline (T1) average diastolic blood pressure - Youth: number analyzed (Participants) | 25 | 17 | 29 | 71
  Baseline (T1) average diastolic blood pressure - Youth | 60.6667 (7.5951) | 64.8431 (6.2607) | 59.954 (6.8503) | 61.3756 (7.1725)
  T2 average diastolic blood pressure - Parents: number analyzed (Participants) | 20 | 16 | 27 | 63
  T2 average diastolic blood pressure - Parents | 68.85 (6.203) | 67.729 (9.092) | 73.0123 (12.8121) | 70.3492 (10.3058)
  T2 average diastolic blood pressure- Youth: number analyzed (Participants) | 20 | 16 | 26 | 62
  T2 average diastolic blood pressure- Youth | 61.850 (8.2266) | 63.4375 (4.3745) | 60.2821 (8.4442) | 61.6022 (7.527)
  T3 average diastolic blood pressure- Parents: number analyzed (Participants) | 15 | 13 | 23 | 51
  T3 average diastolic blood pressure- Parents | 71.3553 (8.8831) | 69.308 (7.7321) | 76.5797 (13.811) | 73.1895 (11.4445)
  T3 average diastolic blood pressure- Youth: number analyzed (Participants) | 14 | 12 | 22 | 48
  T3 average diastolic blood pressure- Youth | 61.0238 (10.2261) | 64.6947 (6.5941) | 59.5152 (5.5394) | 61.2501 (7.5673)

26. Secondary Outcome: Total Cholesterol
Description: Total cholesterol measured via finger prick blood sample. Total cholesterol is measured in milligrams of cholesterol per deciliter of blood. Scores 200 mg/dL and over are considered high.
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Only a small subsample was selected for this additional biometric data collection. Youth data is incomplete due to the fact that their cholesterol levels were too low for the machine to read. In those cases, the machine displayed "LOW," and were not able to be included in the analysis below.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Groups
Number analyzed (Participants) | 212 | 110 | 156 | 478
mg/dL
  Baseline (T1) total cholesterol- Parents: number analyzed (Participants) | 21 | 15 | 23 | 59
  Baseline (T1) total cholesterol- Parents | 205.29 (83.733) | 188 (21.922) | 200.7 (86.173) | 199.1 (73.465)
  Baseline (T1) total cholesterol- Youth: number analyzed (Participants) | 16 | 12 | 15 | 43
  Baseline (T1) total cholesterol- Youth | 163.38 (11.477) | 167.5 (9.298) | 160.27 (1.787) | 163.44 (11.51)
  T2 total cholesterol- Parents: number analyzed (Participants) | 15 | 12 | 17 | 44
  T2 total cholesterol- Parents | 185.267 (31.227) | 178.667 (23.952) | 215.471 (95.568) | 195.136 (63.206)
  T2 total cholesterol- Youth: number analyzed (Participants) | 11 | 6 | 11 | 28
  T2 total cholesterol- Youth | 159.636 (8.2131) | 163.667 (10.328) | 163.364 (9.4369) | 161.964 (9.0205)
  T3 total cholesterol- Parents: number analyzed (Participants) | 8 | 10 | 16 | 34
  T3 total cholesterol- Parents | 195.88 (27.315) | 169.7 (15.392) | 188.13 (30.289) | 184.53 (27.277)
  T3 total cholesterol- Youth: number analyzed (Participants) | 3 | 8 | 10 | 21
  T3 total cholesterol- Youth | 164.33 (10.116) | 158.63 (7.8) | 164.3 (16.826) | 162.14 (12.91)

27. Secondary Outcome: Glycosylated Hemoglobin (HbA1c)
Description: HbA1c measured via finger prick blood sample using a point of care device; this measures the average blood sugar levels over the past 3 months. For people without diabetes, the normal range for the hemoglobin A1c level is between 4% and 5.6%.
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Parents and youth reported separately. Biometric data was collected from a small subset of participants.
Measure: Mean (Standard Deviation); unit: percentage of total hemoglobin
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Groups
Number analyzed (Participants) | 212 | 110 | 156 | 478
percentage of total hemoglobin
  Baseline (T1) HbA1c - Parents: number analyzed (Participants) | 26 | 17 | 29 | 72
  Baseline (T1) HbA1c - Parents | 5.435 (.5614) | 5.759 (1.9497) | 5.679 (1.7214) | 5.61 (1.4679)
  Baseline (T1) HbA1c - Youth: number analyzed (Participants) | 24 | 17 | 27 | 68
  Baseline (T1) HbA1c - Youth | 5.142 (.3911) | 5.212 (.5566) | 4.981 (.3211) | 5.096 (.4195)
  T2 HbA1c - Parents: number analyzed (Participants) | 20 | 16 | 27 | 63
  T2 HbA1c - Parents | 5.715 (.504) | 5.706 (1.9965) | 5.7 (1.546) | 5.706 (1.423)
  T2 HbA1c - Youth: number analyzed (Participants) | 20 | 16 | 25 | 61
  T2 HbA1c - Youth | 5.225 (.3823) | 5.238 (.55) | 5.044 (.4925) | 5.154 (.477)
  T3 HbA1c - Parents: number analyzed (Participants) | 15 | 13 | 23 | 51
  T3 HbA1c - Parents | 5.7 (.594) | 5.577 (.5644) | 6.096 (1.659) | 5.847 (1.2)
  T3 HbA1c - Youth: number analyzed (Participants) | 14 | 12 | 20 | 46
  T3 HbA1c - Youth | 5.521 (.7051) | 5.35 (.2876) | 5.525 (.7538) | 5.478 (.6401)

28. Secondary Outcome: Parent and Adolescent Diet- Total Energy (kcal)
Description: Total energy from food (kcal) based off 24 hour food recalls
Time Frame: Week 0 (t1), Week 10-12 (T2), Week 24-26 (T3)
Population: Only a small subset was selected to participate in these additional data collection measures.
Measure: Mean (Standard Deviation); unit: kcal.
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Groups
Number analyzed (Participants) | 106 | 55 | 78 | 239
kcal.
  Baseline (T1) kcal.- Parents: number analyzed (Participants) | 35 | 17 | 29 | 81
  Baseline (T1) kcal.- Parents | 1450.440 (452.629) | 1594.887 (525.105) | 1394.403 (448.198) | 1460.693 (466.896)
  Baseline (T1) kcal.- Youth: number analyzed (Participants) | 30 | 14 | 27 | 72
  Baseline (T1) kcal.- Youth | 1436.607 (551.683) | 1501.483 (485.299) | 1408.204 (691.582) | 1439.471 (603.163)
  T2 kcal.- Parents: number analyzed (Participants) | 22 | 14 | 24 | 60
  T2 kcal.- Parents | 1282.684 (343.439) | 1264.033 (398.669) | 1396.699 (513.453) | 1323.938 (428.269)
  T2 kcal.- Youth: number analyzed (Participants) | 23 | 14 | 23 | 60
  T2 kcal.- Youth | 1531.126 (506.809) | 1116.894 (485.300) | 1619.568 (552.873) | 1468.375 (549.007)
  T3 kcal.- Parents: number analyzed (Participants) | 19 | 13 | 23 | 55
  T3 kcal.- Parents | 1322.501 (424.671) | 1533.335 (455.535) | 1363.178 (519.757) | 1389.372 (472.378)
  T3 kcal.- Youth: number analyzed (Participants) | 22 | 13 | 22 | 57
  T3 kcal.- Youth | 1556.714 (717.439) | 1412.479 (374.180) | 1434.018 (663.167) | 1476.462 (626.204)

29. Secondary Outcome: Parent and Adolescent Diet- Total Dietary Fiber (g)
Description: Total dietary fiber in grams, based on 24 hour food recalls.
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Only a small subset was selected to participate in these additional data collection measures.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Groups
Number analyzed (Participants) | 106 | 55 | 78 | 239
grams
  Baseline (T1) fiber (g)- Parents: number analyzed (Participants) | 35 | 17 | 29 | 81
  Baseline (T1) fiber (g)- Parents | 17.283 (8.292) | 19.344 (6.462) | 16.811 (9.126) | 17.546 (8.225)
  Baseline (T1) fiber (g)- Youth: number analyzed (Participants) | 30 | 15 | 27 | 72
  Baseline (T1) fiber (g)- Youth | 13.036 (6.995) | 13.382 (7.263) | 11.906 (10.428) | 12.684 (8.402)
  T2 fiber (g) - Parents: number analyzed (Participants) | 22 | 14 | 24 | 60
  T2 fiber (g) - Parents | 19.921 (15.253) | 17.830 (7.440) | 18.023 (8.078) | 18.674 (11.016)
  T2 fiber (g) - Youth: number analyzed (Participants) | 23 | 14 | 23 | 60
  T2 fiber (g) - Youth | 14.469 (7.614) | 9.724 (3.673) | 13.657 (7.595) | 13.050 (7.047)
  T3 fiber (g) - Parents: number analyzed (Participants) | 19 | 13 | 23 | 55
  T3 fiber (g) - Parents | 17.468 (7.464) | 20.589 (8.980) | 16.957 (9.248) | 17.992 (8.574)
  T3 fiber (g) - Youth: number analyzed (Participants) | 22 | 13 | 22 | 57
  T3 fiber (g) - Youth | 15.312 (11.811) | 14.190 (5.485) | 14.835 (9.765) | 14.872 (9.731)

30. Secondary Outcome: Home Food Environment - Vegetable Availability
Description: Modified version of the validated Home Food Inventory with cultural adaptations including foods commonly consumed by Latinos used to inventory number of different vegetable items present in the home. Reporting on variable: # of vegetable items present in the home.
Time Frame: Week 0 (Time 1), Week 10-12 (T2), Week 24-26 (T3)
Population: Only a small subset was selected to participate in these additional data collection measures. T3 is very small due to COVID; home visits were suspended.
Measure: Mean (Standard Deviation); unit: count of vegetables
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Conditions
Number analyzed (Participants) | 106 | 55 | 78 | 239
count of vegetables
  T1 (week 0) count of vegetables in the home: number analyzed (Participants) | 26 | 17 | 29 | 72
  T1 (week 0) count of vegetables in the home | 8.3846 (3.2382) | 8.4706 (3.8587) | 8.931 (3.401) | 8.625 (3.4168)
  T2 (week 10-12) count of vegetables in the home: number analyzed (Participants) | 20 | 16 | 27 | 63
  T2 (week 10-12) count of vegetables in the home | 9.25 (2.9177) | 9.4375 (2.7561) | 8.3333 (3.3050) | 8.9048 (3.0465)
  T3 (week 24-26) count of vegetables in the home: number analyzed (Participants) | 14 | 13 | 24 | 51
  T3 (week 24-26) count of vegetables in the home | 7.5714 (2.8206) | 8.3846 (3.501) | 8.9583 (3.0571) | 8.4314 (3.1065)

31. Secondary Outcome: BMI % for Youth
Description: BMI percentile, expressing a child's BMI relative to US children who participated in national surveys from 1963-65 to 1988-94. Typically, weight status categories are as follows: healthy weight is considered 5th percentile to less than the 85th percentile; 85th to less than the 95th percentile indicates overweight, and above the 95th percentile indicates obesity.
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Only a small subset was selected to participate in these additional biometric data collection measures.
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Groups
Number analyzed (Participants) | 106 | 55 | 78 | 239
percentile
  Baseline (T1) BMI %- Youth: number analyzed (Participants) | 25 | 17 | 29 | 71
  Baseline (T1) BMI %- Youth | 78.512 (21.8731) | 91.8176 (11.996) | 78.3 (21.9048) | 81.6113 (20.5458)
  T2 BMI %- Youth: number analyzed (Participants) | 20 | 16 | 26 | 62
  T2 BMI %- Youth | 80.01 (17.2701) | 91.25 (10.7304) | 76.7885 (23.686) | 81.5597 (19.6535)
  T3 BMI %- Youth: number analyzed (Participants) | 14 | 12 | 22 | 48
  T3 BMI %- Youth | 72.67 (20.304) | 95.73 (4.161) | 76.5 (22.113) | 80.19 (20.53)

32. Secondary Outcome: Parent and Adolescent Diet - % Calories From Fat
Description: Percentage of daily calories that come from fat
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Only a small subset was selected to participate in these additional data collection measures.
Measure: Mean (Standard Deviation); unit: percentage of calories from fat
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Groups
Number analyzed (Participants) | 106 | 55 | 78 | 239
percentage of calories from fat
  Baseline (T1) % calories from fat- Parents: number analyzed (Participants) | 35 | 17 | 29 | 81
  Baseline (T1) % calories from fat- Parents | 34.038 (8.782) | 31.825 (5.385) | 31.315 (9.031) | 32.599 (8.292)
  Baseline (T1) % calories from fat- Youth: number analyzed (Participants) | 30 | 15 | 27 | 72
  Baseline (T1) % calories from fat- Youth | 31.248 (7.053) | 33.789 (6.667) | 34.206 (8.668) | 32.887 (7.653)
  T2 % calories from fat- Parents: number analyzed (Participants) | 22 | 14 | 24 | 60
  T2 % calories from fat- Parents | 30.756 (8.700) | 31.933 (8.189) | 30.408 (6.974) | 30.891 (7.813)
  T2 % calories from fat - Youth: number analyzed (Participants) | 23 | 14 | 23 | 60
  T2 % calories from fat - Youth | 30.091 (7.957) | 29.294 (6.390) | 32.787 (7.768) | 30.939 (7.573)
  T3 % calories from fat- Parents: number analyzed (Participants) | 19 | 13 | 23 | 55
  T3 % calories from fat- Parents | 34.484 (7.412) | 33.087 (8.199) | 31.174 (8.015) | 32.770 (7.846)
  T3 % calories from fat- Youth: number analyzed (Participants) | 22 | 13 | 22 | 57
  T3 % calories from fat- Youth | 34.706 (9.953) | 33.101 (6.822) | 32.476 (5.923) | 33.479 (7.829)

33. Secondary Outcome: Parent and Adolescent Diet - % Calories From Carbs
Description: Percentage of daily calories that come from carbohydrate sources
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Only a small subset was selected to participate in these additional data collection measures.
Measure: Mean (Standard Deviation); unit: percentage of calories from carbs
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Groups
Number analyzed (Participants) | 106 | 55 | 78 | 239
percentage of calories from carbs
  Baseline (T1) % calories from carbs- Parents: number analyzed (Participants) | 35 | 17 | 29 | 81
  Baseline (T1) % calories from carbs- Parents | 45.89 (10.302) | 48.727 (7.914) | 50.131 (9.860) | 48.004 (9.765)
  Baseline (T1) % calories from carbs- Youth: number analyzed (Participants) | 30 | 15 | 27 | 72
  Baseline (T1) % calories from carbs- Youth | 49.802 (7.450) | 49.726 (8.621) | 47.929 (9.354) | 49.084 (8.378)
  T2 % calories from carbs- Parents: number analyzed (Participants) | 22 | 14 | 24 | 60
  T2 % calories from carbs- Parents | 48.787 (9.432) | 47.063 (11.065) | 51.439 (7.512) | 49.479 (9.150)
  T2 % calories from carbs- Youth: number analyzed (Participants) | 23 | 14 | 23 | 60
  T2 % calories from carbs- Youth | 52.069 (8.306) | 53.484 (9.318) | 49.955 (9.391) | 51.589 (8.929)
  T3 % calories from carbs- Parents: number analyzed (Participants) | 19 | 13 | 23 | 55
  T3 % calories from carbs- Parents | 45.763 (10.057) | 45.812 (8.887) | 49.451 (10.898) | 47.317 (10.148)
  T3 % calories from carbs- Youth: number analyzed (Participants) | 22 | 13 | 22 | 57
  T3 % calories from carbs- Youth | 48.062 (9.730) | 51.038 (8.945) | 49.895 (6.651) | 49.448 (8.406)

34. Secondary Outcome: Parent and Adolescent Diet - % Calories From Protein
Description: Percentage of daily calories that come from protein sources
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Only a small subset was selected to participate in these additional data collection measures.
Measure: Mean (Standard Deviation); unit: percentage of calories from protein
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Groups
Number analyzed (Participants) | 106 | 55 | 78 | 239
percentage of calories from protein
  Baseline (T1) % calories from protein- Parents: number analyzed (Participants) | 35 | 17 | 29 | 81
  Baseline (T1) % calories from protein- Parents | 19.725 (5.475) | 19.412 (4.978) | 18.505 (5.107) | 19.223 (5.209)
  Baseline (T1) % calories from protein- Youth: number analyzed (Participants) | 30 | 15 | 27 | 72
  Baseline (T1) % calories from protein- Youth | 18.895 (6.173) | 16.448 (4.142) | 17.817 (5.285) | 17.981 (5.480)
  T2 % calories from protein- Parents: number analyzed (Participants) | 22 | 14 | 24 | 60
  T2 % calories from protein- Parents | 20.385 (5.313) | 20.968 (7.765) | 17.691 (6.061) | 19.443 (6.307)
  T2 % calories from protein- Youth: number analyzed (Participants) | 23 | 14 | 23 | 60
  T2 % calories from protein- Youth | 17.875 (3.581) | 17.195 (4.683) | 17.193 (5.633) | 17.455 (4.643)
  T3 % calories from protein- Parents: number analyzed (Participants) | 19 | 13 | 23 | 55
  T3 % calories from protein- Parents | 19.471 (5.183) | 21.127 (8.045) | 19.191 (6.005) | 19.745 (6.216)
  T3 % calories from protein- Youth: number analyzed (Participants) | 22 | 13 | 22 | 57
  T3 % calories from protein- Youth | 17.235 (3.013) | 15.844 (3.842) | 17.616 (4.434) | 17.065 (3.797)

35. Secondary Outcome: Parent and Adolescent Diet - % Calories From Saturated Fats
Description: Percentage of daily calories that come from saturated fat sources
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Only a small subset was selected to participate in these additional data collection measures.
Measure: Mean (Standard Deviation); unit: percentage of calories from sat. fat
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Groups
Number analyzed (Participants) | 106 | 55 | 78 | 239
percentage of calories from sat. fat
  Baseline (T1) % calories from saturated fat- Parents: number analyzed (Participants) | 35 | 17 | 29 | 81
  Baseline (T1) % calories from saturated fat- Parents | 10.784 (4.401) | 10.867 (2.071) | 10.306 (3.783) | 10.630 (3.763)
  Baseline (T1) % calories from saturated fat- Youth: number analyzed (Participants) | 30 | 15 | 27 | 72
  Baseline (T1) % calories from saturated fat- Youth | 10.697 (2.797) | 11.245 (2.433) | 11.717 (3.038) | 11.193 (2.819)
  T2 % calories from saturated fat- Parents: number analyzed (Participants) | 22 | 14 | 24 | 60
  T2 % calories from saturated fat- Parents | 10.235 (4.001) | 10.397 (2.891) | 10.171 (3.048) | 10.247 (3.342)
  T2 % calories from saturated fat- Youth: number analyzed (Participants) | 23 | 14 | 23 | 60
  T2 % calories from saturated fat- Youth | 9.997 (3.387) | 10.675 (2.658) | 10.242 (3.117) | 10.249 (3.086)
  T3 % calories from saturated fat- Parents: number analyzed (Participants) | 19 | 13 | 23 | 55
  T3 % calories from saturated fat- Parents | 10.602 (2.945) | 10.326 (2.551) | 10.309 (3.436) | 10.414 (3.027)
  T3 % calories from saturated fat- Youth: number analyzed (Participants) | 22 | 13 | 22 | 57
  T3 % calories from saturated fat- Youth | 11.648 (3.106) | 10.753 (2.318) | 10.359 (2.291) | 10.946 (2.660)

36. Secondary Outcome: Parent and Adolescent Diet - % Calories From Monounsaturated Fats
Description: Percentage of daily calories that come from monounsaturated fat sources (MUFA).
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Only a small subset was selected to participate in these additional data collection measures.
Measure: Mean (Standard Deviation); unit: percentage of calories from MUFA
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Groups
Number analyzed (Participants) | 106 | 55 | 78 | 239
percentage of calories from MUFA
  Baseline (T1) % calories from mono fat- Parents: number analyzed (Participants) | 35 | 17 | 29 | 81
  Baseline (T1) % calories from mono fat- Parents | 11.680 (2.894) | 11.363 (2.739) | 10.713 (3.697) | 11.268 (3.167)
  Baseline (T1) % calories from mono fat- Youth: number analyzed (Participants) | 30 | 15 | 27 | 72
  Baseline (T1) % calories from mono fat- Youth | 10.387 (2.707) | 11.023 (2.794) | 11.168 (3.374) | 10.812 (2.973)
  T2 % calories from mono fat- Parents: number analyzed (Participants) | 22 | 14 | 24 | 60
  T2 % calories from mono fat- Parents | 11.026 (3.496) | 11.058 (2.435) | 10.667 (2.678) | 10.890 (2.913)
  T2 % calories from mono fat- Youth: number analyzed (Participants) | 23 | 14 | 23 | 60
  T2 % calories from mono fat- Youth | 9.956 (3.399) | 9.917 (2.802) | 11.143 (2.917) | 10.402 (3.091)
  T3 % calories from mono fat- Parents: number analyzed (Participants) | 19 | 13 | 23 | 55
  T3 % calories from mono fat- Parents | 12.719 (3.350) | 12.095 (4.594) | 11.164 (3.946) | 11.919 (3.904)
  T3 % calories from mono fat- Youth: number analyzed (Participants) | 22 | 13 | 22 | 57
  T3 % calories from mono fat- Youth | 11.667 (3.764) | 11.568 (2.765) | 11.384 (2.550) | 11.535 (3.067)

37. Secondary Outcome: Parent and Adolescent Diet - % Calories From Polyunsaturated Fats
Description: Percentage of daily calories that come from polyunsaturated fat sources (PUFA).
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Only a small subset was selected to participate in these additional data collection measures.
Measure: Mean (Standard Deviation); unit: percentage of calories from PUFA
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Groups
Number analyzed (Participants) | 106 | 55 | 78 | 239
percentage of calories from PUFA
  Baseline (T1) % calories from poly fat- Parents: number analyzed (Participants) | 35 | 17 | 29 | 81
  Baseline (T1) % calories from poly fat- Parents | 8.365 (5.408) | 6.431 (1.739) | 7.244 (3.075) | 7.558 (4.116)
  Baseline (T1) % calories from poly fat- Youth: number analyzed (Participants) | 30 | 15 | 27 | 72
  Baseline (T1) % calories from poly fat- Youth | 7.108 (2.761) | 8.366 (2.857) | 8.185 (3.440) | 7.774 (3.063)
  T2 % calories from poly fat- Parents: number analyzed (Participants) | 22 | 14 | 24 | 60
  T2 % calories from poly fat- Parents | 6.421 (2.203) | 7.183 (4.405) | 6.797 (2.752) | 6.749 (3.007)
  T2 % calories from poly fat- Youth: number analyzed (Participants) | 23 | 14 | 23 | 60
  T2 % calories from poly fat- Youth | 7.218 (3.266) | 6.037 (2.113) | 8.470 (3.083) | 7.423 (3.067)
  T3 % calories from poly fat- Parents: number analyzed (Participants) | 19 | 13 | 23 | 55
  T3 % calories from poly fat- Parents | 7.615 (2.716) | 7.391 (3.298) | 6.655 (1.988) | 7.161 (2.585)
  T3 % calories from poly fat- Youth: number analyzed (Participants) | 22 | 13 | 22 | 57
  T3 % calories from poly fat- Youth | 8.109 (3.597) | 7.797 (2.225) | 7.716 (3.417) | 7.887 (3.213)

38. Secondary Outcome: Parent and Adolescent Diet - Total Sugars (g)
Description: Total sugars in daily diet, measured in grams.
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Only a small subset was selected to participate in these additional data collection measures.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Groups
Number analyzed (Participants) | 106 | 55 | 78 | 239
grams
  Baseline (T1) total sugars (g) - Parents: number analyzed (Participants) | 35 | 17 | 24 | 81
  Baseline (T1) total sugars (g) - Parents | 66.608 (37.864) | 75.698 (33.378) | 69.385 (30.359) | 69.511 (34.154)
  Baseline (T1) total sugars (g) - Youth: number analyzed (Participants) | 30 | 15 | 27 | 72
  Baseline (T1) total sugars (g) - Youth | 78.104 (37.468) | 74.251 (34.586) | 71.425 (41.784) | 74.791 (38.179)
  T2 total sugars (g) - Parents: number analyzed (Participants) | 22 | 14 | 24 | 60
  T2 total sugars (g) - Parents | 64.893 (28.514) | 61.821 (29.546) | 73.491 (41.367) | 67.616 (34.258)
  T2 total sugars (g) - Youth: number analyzed (Participants) | 23 | 14 | 23 | 60
  T2 total sugars (g) - Youth | 84.194 (43.139) | 58.984 (31.743) | 80.593 (28.161) | 76.932 (36.247)
  T3 total sugars (g) - Parents: number analyzed (Participants) | 19 | 13 | 23 | 55
  T3 total sugars (g) - Parents | 56.714 (30.960) | 67.495 (32.236) | 71.231 (35.761) | 65.334 (33.369)
  T3 total sugars (g) - Youth: number analyzed (Participants) | 22 | 13 | 22 | 57
  T3 total sugars (g) - Youth | 6.968 (27.827) | 72.752 (43.290) | 70.566 (40.806) | 69.676 (36.356)

39. Secondary Outcome: Parent and Adolescent Diet - Added Sugars (g)
Description: Total added sugars in daily diet, measured in grams. This does not include foods like fruit, with naturally occurring sugars.
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Only a small subset was selected to participate in these additional data collection measures.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Groups
Number analyzed (Participants) | 106 | 55 | 78 | 239
grams
  Baseline (T1) added sugars (g) - Parents: number analyzed (Participants) | 35 | 17 | 29 | 81
  Baseline (T1) added sugars (g) - Parents | 38.240 (35.049) | 40.129 (27.235) | 44.178 (25.329) | 40.763 (30.034)
  Baseline (T1) added sugars (g) - Youth: number analyzed (Participants) | 30 | 15 | 27 | 72
  Baseline (T1) added sugars (g) - Youth | 36.007 (21.542) | 32.434 (16.921) | 39.429 (31.181) | 36.545 (24.678)
  T2 added sugars (g) - Parents: number analyzed (Participants) | 22 | 14 | 24 | 60
  T2 added sugars (g) - Parents | 33.009 (20.427) | 30.712 (27.694) | 43.909 (28.673) | 36.832 (25.937)
  T2 added sugars (g) - Youth: number analyzed (Participants) | 23 | 14 | 23 | 60
  T2 added sugars (g) - Youth | 40.828 (30.790) | 32.595 (26.912) | 45.323 (22.842) | 40.630 (27.047)
  T3 added sugars (g) - Parents: number analyzed (Participants) | 19 | 13 | 23 | 55
  T3 added sugars (g) - Parents | 29.023 (20.959) | 34.623 (22.056) | 37.632 (25.691) | 33.947 (23.192)
  T3 added sugars (g) - Youth: number analyzed (Participants) | 22 | 13 | 22 | 57
  T3 added sugars (g) - Youth | 32.448 (18.700) | 38.764 (27.712) | 39.752 (31.875) | 36.701 (26.235)

40. Secondary Outcome: Parent and Adolescent Diet - Whole Grains (oz)
Description: Total whole grains in daily diet, measured in ounce equivalents (oz).
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Only a small subset was selected to participate in these additional data collection measures.
Measure: Mean (Standard Deviation); unit: ounces
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Groups
Number analyzed (Participants) | 106 | 55 | 78 | 239
ounces
  Baseline (T1) whole grains (oz) - Parents: number analyzed (Participants) | 35 | 17 | 29 | 81
  Baseline (T1) whole grains (oz) - Parents | 2.393 (1.635) | 3.594 (2.782) | 2.032 (1.807) | 2.516 (2.041)
  Baseline (T1) whole grains (oz) - Youth: number analyzed (Participants) | 30 | 15 | 15 | 72
  Baseline (T1) whole grains (oz) - Youth | 1.691 (1.442) | 1.657 (1.608) | 1.657 (1.608) | 1.472 (1.345)
  T2 whole grains (oz) - Parents: number analyzed (Participants) | 22 | 14 | 24 | 60
  T2 whole grains (oz) - Parents | 2.352 (1.738) | 2.048 (1.531) | 2.913 (1.793) | 2.589 (1.708)
  T2 whole grains (oz) - Youth: number analyzed (Participants) | 23 | 14 | 14 | 60
  T2 whole grains (oz) - Youth | 2.403 (2.442) | 1.395 (1.307) | 1.395 (1.308) | 2.037 (2.120)
  T3 whole grains (oz) - Parents: number analyzed (Participants) | 19 | 13 | 23 | 55
  T3 whole grains (oz) - Parents | 2.645 (1.681) | 3.576 (2.520) | 2.766 (1.842) | 2.916 (1.969)
  T3 whole grains (oz) - Youth: number analyzed (Participants) | 22 | 13 | 13 | 57
  T3 whole grains (oz) - Youth | 1.385 (1.881) | 1.909 (1.201) | 1.909 (1.201) | 1.670 (2.011)

41. Secondary Outcome: Parent and Adolescent Diet - Refined Grains (oz)
Description: Total refined grains in daily diet, measured in ounce equivalents (oz).
Time Frame: Week 0 (T1), Week 10-12 (T2), Week 24-26 (T3)
Population: Only a small subset was selected to participate in these additional data collection measures.
Measure: Mean (Standard Deviation); unit: ounces
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program | All Groups
Number analyzed (Participants) | 106 | 55 | 78 | 239
ounces
  Baseline (T1) refined grains (oz) - Parents: number analyzed (Participants) | 35 | 17 | 29 | 81
  Baseline (T1) refined grains (oz) - Parents | 2.498 (1.901) | 3.578 (2.518) | 3.256 (2.057) | 2.996 (2.119)
  Baseline (T1) refined grains (oz) - Youth: number analyzed (Participants) | 30 | 15 | 27 | 72
  Baseline (T1) refined grains (oz) - Youth | 3.918 (2.369) | 4.959 (2.473) | 4.522 (2726) | 4.361 (2.528)
  T2 refined grains (oz) - Parents: number analyzed (Participants) | 22 | 14 | 24 | 60
  T2 refined grains (oz) - Parents | 2.199 (1.702) | 2.352 (2.213) | 2.853 (1.910) | 2.419 (1.918)
  T2 refined grains (oz) - Youth: number analyzed (Participants) | 23 | 14 | 23 | 60
  T2 refined grains (oz) - Youth | 4.343 (2.213) | 3.677 (3.225) | 4.836 (3.072) | 4.376 (2.799)
  T3 refined grains (oz) - Parents: number analyzed (Participants) | 19 | 13 | 23 | 55
  T3 refined grains (oz) - Parents | 2.351 (1.901) | 2.645 (2.210) | 2.733 (1.992) | 2.580 (1.984)
  T3 refined grains (oz) - Youth: number analyzed (Participants) | 22 | 13 | 22 | 57
  T3 refined grains (oz) - Youth | 4.398 (3.236) | 4.221 (2.255) | 3.962 (2.347) | 4.189 (2.669)

ADVERSE EVENTS:
Time Frame: Adverse event data were monitored and up to the T3 data collection time point (i.e., 24-26 weeks post intervention start) for each cohort of participants.
Arm/Group | Nutrition/Substance Use Prevention | Substance Use Prevention Only | Academic Success Program
All-Cause Mortality (participants affected / at risk) | 0/361 | 0/222 | 0/261
Serious Adverse Events (participants affected / at risk) | 0/361 | 0/222 | 0/261
Other Adverse Events (participants affected / at risk) | 0/361 | 0/222 | 0/261

LIMITATIONS AND CAVEATS:
Enrollment numbers were smaller due to cancellations caused by social distancing restrictions caused by the global pandemic after March of 2020.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT03517111/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/11/NCT03517111/ICF_001.pdf